CLINICAL TRIAL: NCT03517345
Title: Investigating the Effects of Prebiotic Supplementation on Metabolic Effects of Roux-en-Y Gastric Bypass Surgery: A Prospective Randomized Trial
Brief Title: The Metabolic Effects of Prebiotic Supplementation After Roux-en-Y Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fulya Turker, Principle Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 31806
Record Dates: First submitted 2018-02-14; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Bariatric Surgery
Keywords: Bariatric surgery; Prebiotics; gut microbiota; GLP-1; PYY
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic group (Experimental): Given a prebiotic product (inulin + oligofructose; 5 g) mixed with conventional yogurt (100 g) which given as snack, twice a day.
  Interventions: Dietary Supplement: Prebiotic
- Control group (Experimental): Given conventional yogurt (100 g) which given as snack, twice a day.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Prebiotic — Prebiotic (Inulin+Oligofructose) consumed as 10 g/d in yogurt (200 g/d)
  Arms: Prebiotic group
Dietary Supplement: Control — The only yogurt consumed as 200 g/d without prebiotic.
  Arms: Control group

SUMMARY:
In this study, it is aimed to evaluate whether the addition of prebiotics to patients' post-operative diets increases Roux-en-Y Gastric Bypass surgery effects. Half of the participants were randomized prebiotic with conventional yogurt, while the other half were randomized only conventional yogurt as a snack

DETAILED DESCRIPTION:
Following bariatric surgery, positive alterations are observed in gut microbiota, intestinal peptides, and inflammatory cytokines. Previous studies demonstrate that prebiotic use alone in a tolerable dose (which is 10 g/day) among obese, overweight, or diabetic individuals accelerated the weight loss by reducing hunger and food intake. Furthermore, it could also contribute to the improvement of glucose homeostasis by increase postprandial PYY and GLP-1 levels. Prebiotics feeds healthy intestinal bacteria and enhances their positive effects. The present positive effects appear with SCFAs that stimulates PYY and GLP-1 release and produced by fermentation of prebiotics by bacteria. From this point forth, it was hypothesized that post-operative pre-probiotic usage may enhance the effects of Roux-en-Y Gastric Bypass (RYGB). In addition, administration of pre-probiotics following RYGB may be considered as a simple and cheap treatment support, especially for protecting patients with poor medicine compliance against nutritional deficiencies, as well as for diabetic patients whose glucose regulations deteriorate in the long term, and for those who regain weight.

With the result that the effects of prebiotic supplementation on metabolic results of RYGB surgery in this prospective, randomized, controlled study with a duration of 24 weeks were tested.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40kg/m2; perform of other types of bariatric surgery except gastric bypass (i.e. sleeve gastrectomy, adjustable gastric band)

Exclusion Criteria: I

* Administration of antibiotics (other than 1 g ampicillin-sulbactam one hour before surgery), the presence of chronic gastrointestinal, liver or kidney diseases and malignancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-04-22 (Actual); Primary Completion 2014-12-05 (Actual); Study Completion 2015-02-10 (Actual)

PRIMARY OUTCOMES:
Plasma GLP-1 levels changes | 6 months
  Change in baseline GLP-1 levels (pM) at 6th month. Measured by plasma samples.
Plasma PYY levels changes | 6 months
  Change in baseline PYY levels (pg/ml) at 6th month. Measured by plasma samples.

SECONDARY OUTCOMES:
Appetite regulation | 6 months
  Change in baseline appetite at 6th month. Subjective appetite assessed with visual analog scales

OTHER OUTCOMES:
weight changes | 6 months
  Change in baseline weight (kg) measurements at 6th month.
fat mass changes | 6 months
  Change in baseline fat mass (kg) measurements at 6th month.
fat free mass changes | 6 months
  Change in baseline fat free mass (kg) measurements at 6th month.
excess weight loss changes | 6 months
  Change in excess weight loss (%) throughout 6months.
serum glucose changes | 6 months
  Change in serum glucose levels (mg/dl) throughout 6months.
serum insulin changes | 6 months
  Change in serum insulin levels (µU/mL) throughout 6months.

REFERENCES:
- [Derived] Calikoglu F, Barbaros U, Uzum AK, Tutuncu Y, Satman I. The Metabolic Effects of Pre-probiotic Supplementation After Roux-en-Y Gastric Bypass (RYGB) Surgery: a Prospective, Randomized Controlled Study. Obes Surg. 2021 Jan;31(1):215-223. doi: 10.1007/s11695-020-04894-6. Epub 2020 Aug 15. PMID 32803709